CLINICAL TRIAL: NCT02317198
Title: Ticagrelor or Prasugrel Versus Clopidogrel in Elderly Patients With an Acute Coronary Syndrome and a High Bleeding Risk: Optimization of Antiplatelet Treatment in High-risk Elderly
Acronym: POPular AGE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St. Antonius Hospital (Other)
Collaborators: UMC Utrecht (Other); Leiden University Medical Center (Other); Meander Medical Center (Other); Medical Center Alkmaar (Other); Isala (Other); Gelre Hospitals (Other); Gelderse Vallei Hospital (Other); Frisius Medisch Centrum (Other); Rijnstate Hospital (Other)
Responsible Party: Principal Investigator, Jurriën M. ten Berg, MD, PhD, MD, PhD, St. Antonius Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PAACS01
Record Dates: First submitted 2014-10-10; First posted 2014-12-15 (Estimated); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Non-ST-elevation Acute Coronary Syndrome; Unstable Angina; Non-ST-elevation Myocardial Infarction
Keywords: Elderly; P2Y12 inhibitors; clopidogrel; ticagrelor
MeSH Terms: conditions — Angina, Unstable; Non-ST Elevated Myocardial Infarction | interventions — Clopidogrel; Ticagrelor; Prasugrel Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Clopidogrel
  Interventions: Drug: Clopidogrel
- Control (Active Comparator): Ticagrelor/Prasugrel
  Interventions: Drug: Ticagrelor or Prasugrel

INTERVENTIONS:
Drug: Clopidogrel
  Other Names: Plavix; Grepid
  Arms: Intervention
Drug: Ticagrelor or Prasugrel
  Arms: Control

SUMMARY:
A randomized controlled, open label, multicenter trial with 1000 patients aged 70 years and older, presenting with Non-ST-elevation acute coronary syndrome. Patients will be randomized to either clopidogrel or the novel P2Y12 inhibitor (ticagrelor or prasugrel). Patients will be followed for one year for outcomes such as bleeding episode requiring medical intervention and net clinical benefit (all cause mortality, non-fatal myocardial infarction, non-fatal stroke, PLATO major and minor bleeding).

ELIGIBILITY:
Inclusion Criteria:

* At least 70 years of age.
* Hospitalization for NSTEMI or UA < 72 hours

Exclusion Criteria:

* Contraindication to P2Y12 inhibitors i.e. clopidogrel, prasugrel or ticagrelor:
* Unable or unwilling to give informed consent or have a life expectancy of less than one year.
* Having received thrombolytic therapy within the previous 24 hours.
* Severe renal function impairment needing dialysis.
* Confirmed or persistent severe hypertension (Systolic Blood Pressure (SBP) > 180 mmHg and/or Diastolic Blood Pressure (DBP) >110 mmHg) at randomization.
* At increased bleeding risk, at the investigator's opinion, e.g. because of malignancy.
* Cardiogenic shock (SBP ≤ 80mmHg for >30 mins) or Intra-Aortic Balloon Pump (IABP) at the time of screening.
* History of major surgery, severe trauma, fracture or organ biopsy within 90 days prior to randomisation.
* Clinically significant out of range values for platelet count or haemoglobin at screening, in the investigator's opinion.
* ACS under dual antiplatelet therapy, e.g. aspirin with a P2Y12 inhibitor; clopidogrel, prasugrel, ticagrelor.
* Patients with a known CYP2C19 genotype at the time of randomization.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1011 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
occurrence of any bleeding episode requiring medical intervention at 1 year after randomisation | One year
net clinical benefit at 1 year after randomisation | One year
  All cause mortality, non-fatal myocardial infarction, non-fatal stroke, PLATO major and minor bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Jurriën M ten Berg, MD, PhD, Principal Investigator — St. Antonius Hospital
Locations (1):
- St. Antonius hospital, Nieuwegein, Utrecht, Netherlands

REFERENCES:
- [Derived] van den Broek WWA, van Paassen JG, Gimbel ME, Deneer VHM, Ten Berg JM, Vreman RA. Cost-effectiveness of clopidogrel vs. ticagrelor in patients of 70 years or older with non-ST-elevation acute coronary syndrome. Eur Heart J Cardiovasc Pharmacother. 2022 Dec 15;9(1):76-84. doi: 10.1093/ehjcvp/pvac037. PMID 35723240
- [Derived] Gimbel M, Qaderdan K, Willemsen L, Hermanides R, Bergmeijer T, de Vrey E, Heestermans T, Tjon Joe Gin M, Waalewijn R, Hofma S, den Hartog F, Jukema W, von Birgelen C, Voskuil M, Kelder J, Deneer V, Ten Berg J. Clopidogrel versus ticagrelor or prasugrel in patients aged 70 years or older with non-ST-elevation acute coronary syndrome (POPular AGE): the randomised, open-label, non-inferiority trial. Lancet. 2020 Apr 25;395(10233):1374-1381. doi: 10.1016/S0140-6736(20)30325-1. PMID 32334703
- [Derived] Qaderdan K, Ishak M, Heestermans AA, de Vrey E, Jukema JW, Voskuil M, de Boer MJ, van't Hof AW, Groenemeijer BE, Vos GJ, Janssen PW, Bergmeijer TO, Kelder JC, Deneer VH, ten Berg JM. Ticagrelor or prasugrel versus clopidogrel in elderly patients with an acute coronary syndrome: Optimization of antiplatelet treatment in patients 70 years and older--rationale and design of the POPular AGE study. Am Heart J. 2015 Nov;170(5):981-985.e1. doi: 10.1016/j.ahj.2015.07.030. Epub 2015 Aug 4. PMID 26542508